CLINICAL TRIAL: NCT04304625
Title: TRAnexamic Acid for Preventing Blood Loss Following a Cesarean Delivery in Women With Placenta pREVIA: a Multicenter Randomised, Double Blind Placebo Controlled Trial
Brief Title: TRAnexamic Acid for Preventing Blood Loss Following a Cesarean Delivery in Women With Placenta pREVIA
Acronym: TRAAPrevia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2018/64
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; tranexamix acid; placenta previa
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta Previa | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multicenter double-blind randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Double blinding is performed according to current Good Manufacturing Practices (BPF). The packaging and labelling of the experimental drugs are carried out by the PUI of CHU Angers, in accordance with the regulation of the clinical trials in force. PUI of CHU Angers will produce batches of vials (tranexamic acid or placebo according to randomization) according to the model:
  * TXA: 1g - 10ml
  * Placebo: NaCl 0.9% - 10mL
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): After the routine prophylactic IV or IM injection of the uterotonic used in the hospital protocol's -either oxytocin or carbetocin - (as recommended by the 2014 guidelines for prevention and management of postpartum hemorrhage from the CNGOF), the intervention will be the IV administration of a 10-ml blinded ampoule of the study drug (either TXA or placebo according to the randomisation sequence) to the patient within 3 minutes after birth, slowly (over 30-60 seconds), once the cord has been clamped
  Interventions: Drug: Tranexamic Acid / Sodium chloride
- Placebo (Placebo Comparator): After the routine prophylactic IV or IM injection of the uterotonic used in the hospital protocol's -either oxytocin or carbetocin - (as recommended by the 2014 guidelines for prevention and management of postpartum hemorrhage from the CNGOF), the intervention will be the IV administration of a 10-ml blinded ampoule of the study drug (either TXA or placebo according to the randomisation sequence) to the patient within 3 minutes after birth, slowly (over 30-60 seconds), once the cord has been clamped
  Interventions: Drug: Tranexamic Acid / Sodium chloride

INTERVENTIONS:
Drug: Tranexamic Acid / Sodium chloride — After the routine prophylactic IV or IM injection of the uterotonic used in the hospital protocol's -either oxytocin or carbetocin - (as recommended by the 2014 guidelines for prevention and management of postpartum hemorrhage from the CNGOF), the intervention will be the IV administration of a 10-ml blinded ampoule of the study drug (either TXA or placebo according to the randomisation sequence) to the patient within 3 minutes after birth, slowly (over 30-60 seconds), once the cord has been clamped

SUMMARY:
Several randomized, controlled trials, mostly involving women undergoing cesarean delivery, have shown that the prophylactic intravenous administration of 1 g of tranexamic acid after childbirth reduced blood loss. Most were small, single-centre trials with considerable methodologic limitations.

It is important to emphasize that none of these RCTs has included women at increased risk of PPH such as placenta previa, a context in which the prevalence of moderate and severe blood loss is significantly higher and where the magnitude of the effect of TXA may highly differ compared to low risk women

DETAILED DESCRIPTION:
TXA is a promising candidate drug, inexpensive and easy to administer, that can be easily added to the delivery management of women worldwide. Strong evidence that TXA reduces blood transfusion in elective and emergency surgery, outside obstetrics, has been available for many years, whatever the type of surgery (ie cardiac, orthopaedic, hepatic, urological, and vascular surgery). Tranexamic acid was recently shown to reduce bleeding-related mortality among women with postpartum hemorrhage, especially when the drug was administered shortly after delivery. A meta-analysis of data from individual patients including data from patients with trauma and women with postpartum hemorrhage suggested the importance of early treatment.

Several randomized, controlled trials (RCTs), involving women undergoing cesarean delivery, as well have meta-analyses, have shown that the prophylactic intravenous administration of 1 g of tranexamic acid after childbirth reduced blood loss. Most of them were small, single- center trials with considerable methodologic limitations. Thus, no guidelines advocate the use of tranexamic acid to prevent blood loss after cesarean delivery. Moreover, it is important to emphasize that none of these RCTs has included women at increased risk of PPH such as placenta previa, a context in which the prevalence of moderate and severe blood loss is significantly higher and where the magnitude of the effect of TXA may highly differ compared to low risk women.

The aim of our study is to conduct a large multicentre randomised, double blind placebo controlled trial to adequately assess the impact of TXA for preventing PPH following a cesarean delivery in women with placenta previa.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years
* Placenta previa defined by a placental edge below 20mm from internal cervical os diagnosed at the most recent transvaginal ultrasound examination before delivery, as per French guidelines
* Cesarean delivery before or during labor
* Gestational age at delivery ≥ 32 weeks + 0
* Affiliated or beneficiary to a health security system
* Signed informed consent

Exclusion Criteria:

* History of venous (deep vein thrombosis and/or pulmonary embolism) or arterial (angina pectoris, myocardial infarction, stroke) thrombotic event
* History of epilepsy or seizure
* Chronic or acute cardiovascular disease (including foramen oval, mitral stenosis, aortic stenosis, heart transplant, pulmonary hypertension); chronic or acute renal disease (including chronic or acute kidney failure with glomerular filtration rate <90 mL/min, renal transplantation), chronic active or acute liver disorder with hemorrhagic or thrombotic risk (including cirrhosis, portal hypertension, Budd-Chiari syndrome)
* Active autoimmune disease with thromboembolic risk (including lupus, antiphospholipid syndrome, Crohn's disease)
* Sickle cell disease (homozygous)
* Severe hemostasis disorder prothrombotic (Factor V Leiden mutation - homo or heterozygous; Activated protein C (APC) resistance, Protein C deficiency, Protein S deficiency - aside from pregnancy, Homocysteinemia, , Factor 2 mutation - homo or heterozygous, Deficiency in antithrombin 3), prohemorragic (von Willebrand disease requiring desmopressin treatment during delivery, thrombocytopenia (<30000/mm3), Glanzmann disease, hypofibrinogenemia (<1g/L) -aside from pregnancy)
* High prenatal suspicion of placenta accreta spectrum disorder according to the obstetrician in charge
* Placenta praevia diagnosed during delivery
* Abruptio placentae
* Significant bleeding (estimated blood loss>500ml) within 12 hours before cesarean delivery
* Eclampsia / HELLP syndrome
* In utero fetal death
* Administration of low-molecular-weight heparin or antiplatelet agents during the 7 days before delivery
* Tranexamic acid contraindication
* Sodium chloride contraindication
* Women under legal protection
* Poor understanding of the French language

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of red blood cell transfusion (binary outcome) between delivery of child and discharge from postpartum hospital stay. | baseline
  Incidence of red blood cell transfusion (binary outcome) between delivery of child and discharge from postpartum hospital stay.

SECONDARY OUTCOMES:
gravimetrically estimated blood loss | Baseline
  gravimetrically estimated blood loss by measuring the suction volume and swab weight (estimated blood loss = (weight of materials used + materials not used - weight of all materials before surgery)/1.05 + volume included in the suction container)
Occurrence of calculated blood loss > 1000ml. | Baseline
  Calculated blood loss = estimated blood volume × (preoperative Ht - postoperative Ht)/preoperative Ht (where estimated blood volume = weight (kg) × 85). Preoperative Ht will be the most recent Ht within 7 days before delivery. Postoperative Ht will be measured at day 2 postpartum
Occurrence of calculated blood loss > 1500ml. | Baseline
  calculated blood loss > 1500 ml
mean calculated blood loss | Baseline
  mean calculated blood loss
linically significant PPH | Baseline
  provider-assessed clinically significant PPH
shock index | 15, 30, 45, 60 and 120 minutes after birth
  mean shock index defined by the ratio of heart rate to systolic blood pressure
supplementary uterotonic treatment | Baseline
  supplementary uterotonic treatment
iron sucrose perfusion | Baseline
  iron sucrose perfusion until discharge
red blood cell units transfusion | Baseline
  number of red blood cell units transfused between delivery of child and discharge from postpartum hospital stay.
number of transfusion | Baseline
  proportion of women transfused between delivery of child and 24 hours postpartum
arterial embolisation | Baseline
  arterial embolisation or emergency surgery for PPH
maternal postpartum transfer | Baseline
  maternal postpartum transfer to a higher level of care
change in peripartum Hb | day 2
  mean change in peripartum Hb (difference between most recent Hb within 7 days before surgery and at day 2 postpartum).
change in peripartum Ht | day 2
  mean change in peripartum Ht (difference between most recent Ht within 7 days before surgery and at day 2 postpartum).
proportion of breastfeeding at hospital discharge | Baseline
  proportion of breastfeeding at hospital discharge
maternal death for any cause | Baseline
  maternal death for any cause
mild adverse reactions of TXA | Hospitalization stay
  mild adverse reactions of TXA for women (e.g.: nausea, vomiting, phosphenes, dizziness)
thromboembolic events | week 12
  Occurrence of thromboembolic events and other severe unexpected adverse reactions (e.g incidence of deep vein thrombosis confirmed by radiological exams, pulmonary embolism confirmed by radiological exams, myocardial infarction, seizure, renal failure necessitating dialysis)
transfer to neonatal ICU | Baseline
  neonatal outcomes: transfer to neonatal ICU
Women's satisfaction and psychological status | Week 8; Week 12
  Women's satisfaction and psychological status (self-administered questionnaire at day 2 postpartum and self-administered questionnaire sent by mail at 8 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sentilhes L, Madar H, Ifrah A, Chretien JM, Deneux-Tharaux C; TRAAPREVIA Study Group, the Groupe de Recherche en Obstetrique et Gynecologie (GROG). Study protocol. TRAAPREVIA-TRAnexamic acid for preventing blood loss following a cesarean delivery in women with a placenta pREVIA or low-lying placenta: a multicenter randomized, double blind, placebo controlled trial. BMC Pregnancy Childbirth. 2025 May 30;25(1):635. doi: 10.1186/s12884-025-07682-1. PMID 40448004
- [Derived] Larson NJ, Mergoum AM, Dries DJ, Cook A, Blondeau B, Rogers FB. THE ROLE OF TRANEXAMIC ACID IN POSTPARTUM HEMORRHAGE: A NARRATIVE REVIEW. Shock. 2024 Nov 1;62(5):620-627. doi: 10.1097/SHK.0000000000002455. Epub 2024 Aug 20. PMID 39162220